CLINICAL TRIAL: NCT05670262
Title: The Roles of Human Microbiome and Vitamin D in the Development of Childhood Allergic Diseases
Status: Recruiting | Type: Observational
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CMUH111-REC2-033
Record Dates: First submitted 2023-01-02; First posted 2023-01-04 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Pediatric
Keywords: allergic diseases; birth cohort; human microbiome; vitamin D; vitamin D receptors and vitamin D binding protein

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A birth cohort study to evaluate the role of human microbiome and vitamin D in the development of allergic diseases in young child before one year of age.

DETAILED DESCRIPTION:
Allergic diseases are chronic inflammatory disorders that frequently affect young infants before one year of age, and is the beginning of allergy march in later life. The prevalence is increasing in industrial world, Taiwan included. Genetic and environmental factors, such exposure to allergens and microbes, especially early in life, have a detrimental role in the development of allergic diseases, such as atopic dermatitis (AD), allergic rhinitis and asthma. Vitamin D has an important role in different allergic disease. Lower cord blood vitamin D status was observed in infants that developed eczema. Vitamin D binding protein (DBP) bound to vitamin D and regulated its metabolites in the circulation. Moreover, vitamin D receptors have been identified on nearly all cells of the immune system. It may contribute to maintenance of intestinal barrier function by preventing increased intestinal permeability, dysbiosis, inflammation, and a lack of immune tolerance in the gut.

Although aberrant interactions between gut microbes and the intestinal immune system have been implicated in this allergic disease, however, the causal effect of microbiota colonization of the gut and vitamin D that influence the development of allergic diseases, such as AD, in young infants is still unknown. The investigators plan to design a birth cohort study to evaluate the role of human microbiome and vitamin D in the development of allergic diseases in young child before one year of age.

In this study, the investigators will recruit mother-infant pairs in antenatal clinics in China Medical University Hospital and China Medical University Children's Hospital. Newborns who have been enrolled at birth are collected for meconium samples before discharged from nursery and eligible for follow-up visits, and collect their nasal and anal swab microbiome samples at 2 and 12 months follow-up visit. Parental questionnaires are collected at 6, and 12 months of age. All infants were assessed at birth, 2 and 6, and 12 months of age. Assessment included physical examination for allergic diseases. In addition, infants at 12 months of age were collected their 3cc of blood sample.

The investigators believe this longitudinal and prospective study, to follow-up infants from the date of birth until one years old, can answer the cause-effect relationships of microbiota and vitamin D in the development of allergic diseases, and design a microbiota-related preventive and treatment strategy.

ELIGIBILITY:
Inclusion Criteria:

* All term newborn babies who are born in China Medical University Hospital. The term baby defines the maternal gestational age between 37 0/7 weeks to 41 6/7 weeks.

Exclusion Criteria:

* The exclusion criteria are prematurity newborn, congenital anomalies and cardiopulmonary failure need for resuscitation immediately after birth.

Ages: 0 Years to 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All term newborn babies who are born in China Medical University Hospital. The term baby defines the maternal gestational age between 37 0/7 weeks to 41 6/7 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2022-08-04 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Microbiome | Month 0
  Meconium samples will be used to detect intestinal microbiome by using 16S rRNA sequencing to determine baseline status.
Microbiome | Month 2
  Nasal and anal swabs will be used to detect respiratory and intestinal microbiome by using 16S rRNA sequencing to determine baseline status.
Microbiome | Month 12
  Nasal and anal swabs will be used to detect respiratory and intestinal microbiome by using 16S rRNA sequencing,and to follow the change from baseline in microbiome at month 12.
Levels of vitamin D | Month 12
  Vitamin D will be measured in a blood sample by ELISA.
Single nucleotide polymorphism of vitamin D receptor and vitamin D binding protein | Month 12
  Single nucleotide polymorphism (SNP) genotyping will be performed in a blood sample by using TaqMan SNP genotyping assays.
Total immunoglobulin E (IgE) | Month 12
  Plasma total IgE concentration will be measured by microparticle immunoassay (IMx analyzer, Abbott Laboratories, Abbott Park, IL) and ELISA.
Allergen-specific immunoglobulin E (IgE) | Month 12
  Plasma allergen-specific IgE will be measured by BioIC ®.

SECONDARY OUTCOMES:
Parental questionnaire (0-6 month) | Month 6
  For assessing child's health, feeding habit, and environmental exposure
Parental questionnaire (6-12 month) | Month 12
  For assessing child's health, feeding habit, and environmental exposure

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan